CLINICAL TRIAL: NCT02391311
Title: Speed of Processing Training With Transcranial Direct Current Stimulation in Older HIV+ Adults (HtDCS)
Brief Title: A Novel Neurorehabilitation Approach for Cognitive Aging With HIV
Acronym: HtDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pariya L. Fazeli, PhD, Principal investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K99AG048762 (NIH)
Record Dates: First submitted 2015-03-05; First posted 2015-03-18 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: HIV; Aging
Keywords: tDCS; Cognitive remediation therapy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham tDCS + Cognitive Remediation (Active Comparator): Subjects in the sham arm will be administered sham transcranial direct current stimulation (tDCS) (i.e., tDCS will be administered for 30 seconds and then will automatically turn off). Sham group will have identical intervention of engagement in 10 1-hour computerized cognitive remediation therapy sessions during sham tDCS as with the active tDCS condition.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Active tDCS + Cognitive Remediation (Experimental): Subjects in the active arm will be administered active transcranial direct current stimulation (tDCS) (i.e., 2.0 mA tDCS will be administered for 20 minutes and then will automatically turn off). Active group will have identical intervention engagement in 10 1-hour computerized cognitive remediation therapy sessions during active tDCS as with the sham tDCS condition.
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS is a low level electrical stimulation that will be applied to F10. The sham group will receive 2 mA (milliamps) for 30 seconds, while the experimental group will receive 2 mA for 20 minutes. Both groups will have 10, 1 hour sessions of playing cognitive remediation games, while receiving the respective level of tDCS for sham vs experimental conditions.
  Other Names: transcranial electrical stimulation (tES)

SUMMARY:
The goal of this study is to conduct a small, self-contained project to test the hypothesis that tDCS will augment SOP cognitive remediation therapy (CRT) in older HIV+ adults. The investigators will randomly assign 60 HIV+ older adults (i.e., ≥ 50 years old) to 10-hours in either a SOP CRT + sham tDCS condition (n=30) or SOP CRT + active tDCS condition (n=30) and examine neurocognitive functioning at baseline and 6 weeks post-intervention. Hypothesis 1: The SOP CRT + active tDCS condition will show larger proximal (i.e., SOP) gains than the SOP CRT + sham tDCS condition. Hypothesis 2: The active tDCS condition will demonstrate generalization to secondary neurocognitive domains compared to the sham tDCS condition.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Aged 50 and older
* Patient at University HIV/AIDS Clinic

Exclusion Criteria:

* Not homeless
* Not blind or deaf
* No significant neuromedical issues (e.g., schizophrenia, bipolar disorder, stroke, epilepsy or history of seizures)
* No pacemaker or other biomedical devices or metal implants
* No untreated hypertension
* Not undergoing chemo or radiation
* No head injury with LOC greater than 30 mins

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pariya L Fazeli, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB 1917 Clinic, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: March 2015, Primary Completion Date: January 2016 and Study Completion Date: January 2016. Recruitment location: University of Alabama at Birmingham.
Pre-assignment Details: 48 subjects were screened/eligible, however the phone screen did not include consenting. 42 showed up for baseline testing and were consented, thus 42 subjects were enrolled. 42 were randomized immediately after baseline testing, however 5 were either lost to followup or deemed ineligible after baseline testing. See below for further breakdown.
Period: Overall Study
Arm/Group | Sham tDCS + Cognitive Remediation | Active tDCS + Cognitive Remediation
Started | 21 | 21
Completed | 18 | 19
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — deemed ineligible after baseline | 1 | 1

BASELINE CHARACTERISTICS:
Population: n=33 subjects were included in final analyses. Of the 37 that completed the study, 4 were deemed ineligible after they had completed the study due to confirmation with medical records they had conditions that may affect neurocognition (stroke and schizophrenia) although they self reported on the screen they did not have these conditions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS + Cognitive Remediation | Active tDCS + Cognitive Remediation | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Full Range); unit: years] | 55.63 [51 to 71] | 56 [52 to 63] | 55.82 [51 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in the Processing of Speed
Description: Computerized and paper & pencil processing speed measures were used to evaluate this outcome. The Letter and Pattern Comparison Tasks are traditional paper and pencil (SOP) measures. Specifically, they assess perceptual speed. In Letter Comparison subjects are shown three sets of 32 pairs of letters containing 3, 6, or 9 segments. The participants are instructed to decide whether the patterns between the pairs are the same or different within each set, with a time limit of 20 sec per set. Pattern Comparison also presents three sets of 32 pairs of patterns with 3, 6, or 9 line segments. Similarly, participants are instructed to decide whether the patterns are the same or different within the 20 sec time limit. For each measure, the total score is the number of correct answers from all three sets. Larger scores indicate better reasoning and cognitive functioning. In this study scores from Letter and Pattern Comparison were combined for a total Letter/Pattern Score.
Time Frame: baseline, 6 week posttest
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sham tDCS + Cognitive Remediation | Active tDCS + Cognitive Remediation
Number analyzed (Participants) | 16 | 17
units on a scale | 2.63 [-7.0 to 12.0] | 6.06 [-6.0 to 23]

2. Secondary Outcome: Change in Driving Simulator Performance
Description: Driving Simulator Performance: Center lane crossings (a count of how many times an individual crosses the centerline during the entire simulator drive). A difference score was taken between time 2 and time 1 and compared between treatment groups (sham condition and tDCS condition). A negative difference score indicates that fewer center line crossings were made at time 2 than time 1, while positive difference scores indicate the opposite direction, and scores of 0 represent no change.
Time Frame: baseline, 6 week posttest
Population: While n=33 was the final sample used for the primary outcome analyses, n=30 was used for the secondary outcome as 3 subjects did not have available simulator data.
Measure: Mean (95% Confidence Interval); unit: Times crossing center lane
Arm/Group | Sham tDCS + Cognitive Remediation | Active tDCS + Cognitive Remediation
Number analyzed (Participants) | 15 | 15
Times crossing center lane | 1.867 [-2.00 to 11.00] | -1.800 [-12.00 to 3.00]

ADVERSE EVENTS:
Time Frame: Functioning at baseline and 6 weeks post-intervention
Arm/Group | Sham tDCS + Cognitive Remediation | Active tDCS + Cognitive Remediation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No